CLINICAL TRIAL: NCT02160574
Title: A 21-Day Evaluation of the Cumulative Irritation Potential of Topically Applied ZuraPrep™ and ZuraPrep™ Without IPA in Healthy Adult Volunteers
Brief Title: Safety Study to Evaluate the Cumulative Irritation Potential of Topically Applied ZuraPrep™ and ZuraPrep™ Without IPA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zurex Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double
Other Study IDs: 130820-302 (ZX-ZP-0017)
Record Dates: First submitted 2014-06-05; First posted 2014-06-10 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-10

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — chlorhexidine gluconate; Sodium Dodecyl Sulfate; citrate, isopropyl alcohol, methylene blue, parabens drug combination; Ethanol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- ZuraPrep (Active Comparator): ZuraPrep will be compared statistically to ZuraPrep without IPA and both to the Positive Control (0.1% Sodium Lauryl Sulfate). The degree of skin irritation caused by the Reference Product (ChloraPrep) and the Negative Control (0.9% Physiological Saline) will be graded.
  Interventions: Drug: ChloraPrep; Drug: 0.1% Sodium Lauryl Sulfate; Drug: 0.9% Physiological Saline; Other: ZuraPrep without IPA

INTERVENTIONS:
Drug: ChloraPrep — The degree of skin irritation caused by ChloraPrep will be graded and compared to ZuraPrep and ZuraPrep without IPA.
  Other Names: Reference Product; 2% Chlorhexidine Gluconate and 70% IPA
Drug: 0.1% Sodium Lauryl Sulfate — The degree of skin irritation caused by 0.1% Sodium Lauryl Sulfate will be graded and compared to ZuraPrep and ZuraPrep without IPA.
  Other Names: Positive Control
Drug: 0.9% Physiological Saline — The degree of skin irritation caused by 0.9% Physiological Saline will be graded and compared to ZuraPrep and ZuraPrep without IPA.
  Other Names: Negative Control
Other: ZuraPrep without IPA — Results from exposure to ZuraPrep will be compared statistically those from exposure to ZuraPrep without IPA
  Other Names: ZuraPrep without Isopropol Alcohol (IPA)

SUMMARY:
This is a safety study to determine the cumulative skin irritation potential of ZuraPrep™ and ZuraPrep™ without Isopropyl Alcohol after repetitive patch applications to skin of human subjects.

DETAILED DESCRIPTION:
This cumulative irritation evaluation is designed to determine the skin irritation potential of ZuraPrep™ and ZuraPrep™ without Isopropyl Alcohol (IPA) after repetitive patch application to skin of healthy human subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects may be of either sex, at least 18 years of age and of any race
* Subjects must be free of tattoos, sunburn, dermatoses, cuts, lesions or other disorders of the skin of the back.
* Subjects must be in good general health

Exclusion Criteria:

* Known allergies to latex, metals, tape and/or adhesives, soap, citric acid, methylene blue, methylparaben, propylparaben, chlorhexidine gluconate, isopropyl alcohol, and sodium lauryl sulfate.
* Exposure of the back region to antimicrobial agents, medicated soaps, medicated shampoos, medicated lotions, strong detergents, sun-tanning, use of tanning beds, or swimming or soaking in pools or hot tubs, in the 7 days prior to, or during the 3-week test period.
* Use of topical or systemic corticosteroid, antihistamine, or anti-inflammatory medications in the 7 days prior to, or during the 3-week test period.
* Current or recent severe illness such as asthma, diabetes, hepatitis, organ transplant, mitral valve prolapse, congenital heart disease, internal prostheses, or any immunocompromised condition such as AIDS or HIV positive.
* Pregnancy, plans to become pregnant, breast-feeding
* Any active skin rash or breaks in the skin of the back
* Any sunburn or tattoos on the skin of the back
* Current active skin disease or inflammatory skin condition including contact dermatitis
* Participation in a clinical study in the past 7 days or current participation in another clinical study
* Any medical condition or use of any medications that, in the opinion of the Principal Investigator, would preclude participation
* Unwillingness to fulfill the performance requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Scoring Scale (0-7) for Visual Evaluation of Skin Condition | 0-21 days post dose
  Results from skin scores of ZuraPrep and ZuraPrep without IPA will be compared statistically, and both will be compared to the Positive Control (0.1% Sodium Lauryl Sulfate).

SECONDARY OUTCOMES:
Scoring Scale (0-7) for Visual Evaluation of Skin Condition | 0-21 days post dose
  The degree of skin irritation caused by the Reference Product (ChloraPrep) and the Negative Control (0.9% Physiological Saline) will be graded.

CONTACTS AND LOCATIONS:
Overall Officials: Esther Campbell, Principal Investigator — BioScience Laboratories, Inc.
Locations (1):
- BioScience Laboratories, Bozeman, Montana, United States